CLINICAL TRIAL: NCT06279923
Title: Clinical Study of Targeting CD19-BAFF CAR-T Cells in the Treatment of Autoimmune Diseases
Brief Title: CD19-BAFF CAR-T Cells Therapy for Patients With Autoimmune Diseases
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Clinical Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TXB2023023
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Autoimmune Diseases
Keywords: CD19-BAFF CAR-T
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of CD19-BAFF Targeted CAR T-cells (Experimental): Dose escalation follows the standard 3+3 dose escalation design. A total of 3 dose levels are set for subjects.
  Interventions: Biological: CD19-BAFF Targeted CAR T-cells

INTERVENTIONS:
Biological: CD19-BAFF Targeted CAR T-cells — Each subject receive CD19-BAFF Targeted CAR T-cells by intravenous infusion
  Other Names: CD19-BAFF Targeted CAR T-cells injection

SUMMARY:
Clinical Trial for the safety and efficacy of CD19-BAFF CAR-T cells therapy for Autoimmune Diseases.

DETAILED DESCRIPTION:
In this study, 45 patients with Autoimmune Diseases include Systemic Lupus Erythematosus、Systemic sclerosis、Dermatomyositis、Immune nephritis and Neuromyelitis optica were proposed to undergo CD19-BAFF CAR-T cell therapy. Under the premise that its safety has been clarified in previous studies, further observation and evaluation of the effectiveness of CD19-BAFF CAR-T cell therapy for Autoimmune Diseases; At the same time, on the basis of expanding the sample size, more safety data on CD19-BAFF CAR-T cell treatment for Autoimmune Diseases were accumulated, including rare and delayed complications.

ELIGIBILITY:
Inclusion Criteria:

* 1. Gender unlimited，18<Age;
* 2. Diagnosed as Autoimmune Diseases（Systemic Lupus Erythematosus，Immune nephritis, Systemic sclerosis，Dermatomyositis，Neuromyelitis optica）and after routine treatment (using more than 2 types drugs, such as hormones and Immunosuppressants，Immunomodulator or Biological agents) are ineffective for more than 6 months or reappear with disease activity and/or no effective treatment after disease remission
* 3. Estimated life expectancy of minimum of 12 weeks;
* 4. The blood routine meets the following standards:

  1. Lymphocyte count>0.3×10e9/L;
  2. Neutrophils ≥0.5×10e9/L;
  3. Hemoglobin ≥60g/L;
  4. Platelet ≥30×10e9/L
* 5. Pregnant/lactating women, or male or female patients who have fertility and are willing to take effective contraceptive measures at least 6 months after the last cell infusion during the study period;
* 6.Those who voluntarily participated in this trial and provided informed consent;

Exclusion Criteria:

* 1. History of craniocerebral trauma, conscious disturbance, epilepsy, cerebrovascular ischemia, and cerebrovascular hemorrhagic diseases;
* 2. Electrocardiogram shows prolonged QT interval, severe heart diseases such as severe arrhythmia in the past;
* 3.Pregnant or lactating women (the safety of this therapy for unborn children is still unknown)
* 4. Patients with HIV infection
* 5. Active infection of hepatitis B virus or hepatitis C virus;
* 6. The proiferation rate is less than 5 times response to CD3/CD28 co-stimulation signal;
* 7. Creatinine>176.8 umol/L, or ALT / AST > 3 times of normal amounts, or bilirubin>51 umol/L;
* 8. Any unsuitable to participate in this trial judged by the investigator;
* 9. Individuals who have received CAR-T therapy, CAR-NK therapy, or any other gene modified cell therapy product within 3 months;
* 10. Received immunosuppressive therapy within one week prior to mononuclear cell collection；
* 11. ndividuals who have used systemic steroid drugs exceeding 20mg/d of prednisone or equivalent doses within one week prior to treatment (excluding those who have recently or are currently using inhaled steroids)；
* 12. Any situation that researchers believe may increase the risk to the subjects or interfere with the trial results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Up to 28 years after Treatment
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | Up to 2 years after Treatment
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
Multiple Myeloma (MM), Overall response rate (ORR) | Up to 2 years after Treatment
  Assessment of ORR (ORR = sCR+CR+VGPR+PR+MR)
Progression-free survival (PFS) | Up to 2 years after Treatment
  The time from randomization or start of study treatment until objective tumor progression or death
Duration of remission,DOR | Up to 1 years after Treatment
  The time from CR/CRi and PR to disease relapsed or death due to disease

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, MD, Principal Investigator — Zhejiang University
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China